CLINICAL TRIAL: NCT01679613
Title: Relative Bioavailability of Nintedanib Given Alone and in Combination With Ketoconazole at Steady State in Healthy Male Volunteers (an Open-label, Randomised, Two-way Cross-over Clinical Phase I Study)
Brief Title: Investigation of Drug-drug Interaction of Nintedanib and Ketoconazole in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1199.161; 2012-001009-26 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-09-03; First posted 2012-09-06 (Estimated); Results first posted 2014-11-27 (Estimated); Last update posted 2014-11-27 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
MeSH Terms: interventions — nintedanib; Ketoconazole

ARMS (4):
- 1 Nintedanib (Reference) (Experimental): single dose, oral with 240 ml water
  Interventions: Drug: Nintedanib
- 2 Nintedanib + Ketoconazole (Test) (Experimental): Nintedanib single dose, Ketoconazole steady state, oral with 240 ml water
  Interventions: Drug: Ketoconazole; Drug: Nintedanib
- 3 Nintedanib (Reference) (Experimental): single dose, oral with 240 ml water
  Interventions: Drug: Nintedanib
- 4 Nintedanib + Ketoconazole (Test) (Experimental): Nintedanib single dose, Ketoconazole steady state, oral with 240 ml water
  Interventions: Drug: Nintedanib; Drug: Ketoconazole

INTERVENTIONS:
Drug: Nintedanib — low or medium dose depending on pilot part
  Arms: 3 Nintedanib (Reference)
Drug: Nintedanib — low dose oral administration
  Arms: 1 Nintedanib (Reference)
Drug: Ketoconazole — oral administration
  Arms: 2 Nintedanib + Ketoconazole (Test)
Drug: Nintedanib — low dose oral administration
  Arms: 2 Nintedanib + Ketoconazole (Test)
Drug: Nintedanib — low or medium dose depending on pilot part
  Arms: 4 Nintedanib + Ketoconazole (Test)
Drug: Ketoconazole — oral administration
  Arms: 4 Nintedanib + Ketoconazole (Test)

SUMMARY:
The objective of the current study is to investigate the relative bioavailability of a single dose of nintedanib low or high dose with and without coadministration of ketoconazole at steady state

ELIGIBILITY:
Inclusion criteria:

1. healthy male subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1199.161.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

REFERENCES:
- [Derived] Luedtke D, Marzin K, Jungnik A, von Wangenheim U, Dallinger C. Effects of Ketoconazole and Rifampicin on the Pharmacokinetics of Nintedanib in Healthy Subjects. Eur J Drug Metab Pharmacokinet. 2018 Oct;43(5):533-541. doi: 10.1007/s13318-018-0467-9. PMID 29500603

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomised, open-label trial with a 2-way cross-over Pilot part, followed by a 2-way cross-over Main part. Subjects participated either in the Pilot part with 2 treatment sequences (A_B and B_A) or in the Main part with treatment sequences (C_D and D_C) with wash-out period of at least 14 days between each sequence.
Groups:
- Nintedanib (Pilot Part)/ Nintedanib+Ketoconazole (Pilot Part): Nintedanib 50mg was given as a single dose (Treatment A). Following a wash out period of at least 14 days, ketoconazole 400mg was given once daily for three days and nintedanib 50 mg was given as a single dose 1 hour (h) after the ketoconazole administration with ketoconazole under steady-state conditions (Treatment B)
- Nintedanib+Ketoconazole (Pilot Part)/ Nintedanib (Pilot Part): Ketoconazole 400mg was given once daily for three days and nintedanib 50 mg was given as a single dose 1 hour (h) after the ketoconazole administration with ketoconazole under steady-state conditions (Treatment B). Following a wash out period of at least 14 days, nintedanib 50mg was given as a single dose (Treatment A).
- Nintedanib (Main Part)/ Nintedanib+Ketoconazole (Main Part): Based on the results from the Pilot part, nintedanib 50mg was given as a single dose (Treatment C). Following a wash out period of at least 14 days, ketoconazole 400mg was given once daily for 3 days followed by administration of nintedanib 50mg as a single dose 1h after administration of ketoconazole, based on the results from the Pilot part. Nintedanib administration was done under steady state ketoconazole (Treatment D)
- Nintedanib+Ketoconazole (Main Part)/ Nintedanib (Main Part): Ketoconazole 400mg was given once daily for 3 days followed by administration of nintedanib 50mg as a single dose 1h after administration of ketoconazole, based on the results from the Pilot part. Nintedanib administration was done under steady state ketoconazole (Treatment D). Following a wash out period of at least 14 days, nintedanib 50mg was given as a single dose, based on the results from the Pilot part (Treatment C).
Period: Overall Study
Arm/Group | Nintedanib (Pilot Part)/ Nintedanib+Ketoconazole (Pilot Part) | Nintedanib+Ketoconazole (Pilot Part)/ Nintedanib (Pilot Part) | Nintedanib (Main Part)/ Nintedanib+Ketoconazole (Main Part) | Nintedanib+Ketoconazole (Main Part)/ Nintedanib (Main Part)
Started | 4 | 4 | 13 | 13
Received Nintedanib (Pilot) | 4 | 3 | 0 | 0
Received Nintedanib+Ketoconazole (Pilot) | 4 | 4 (One subject received only ketoconazole not nintedanib) | 0 | 0
Received Nintedanib (Main) | 0 | 0 | 13 | 11
Received Nintedanib+Ketoconazole (Main) | 0 | 0 | 13 (Two subjects received only ketoconazole not nintedanib) | 13 (Two subjects received only ketoconazole not nintedanib)
Completed | 4 | 3 | 11 | 11
Not Completed | 0 | 1 | 2 | 2
Not completed — other than stated above | 0 | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Population: The treated set (TS) includes all subjects who were dispensed study medication and were documented to have taken at least one dose of study medication (nintedanib or ketoconazole).
Groups:
- Overall Study: This was a randomised, open-label trial in healthy male subjects with a 2-way cross-over Pilot part, followed by a 2-way cross-over Main part. Subjects participated either in the Pilot part with 2 treatments (A and B) given in 1 of the 2 treatment sequences (A_B and B_A) or in the Main part with also 2 treatments (C and D) given in 1 of the 2 treatment sequences (C_D and D_C). Nintedanib administrations of the 2 respective treatments (A and B or C and D) were to be separated by a wash-out period of at least 14 days. The Pilot part was separated from the Main part by at least 3 weeks to allow for interim analysis
Arm/Group | Overall Study
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 34

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From 0 Extrapolated to Infinity (AUC0-∞)
Description: AUC0-∞ represents the Area under the concentration-time curve of nintedanib in plasma over the time interval from 0 extrapolated to infinity
  For this endpoint, the "measured values" show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities
Time Frame: 1 hour (h) before drug administration and 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 6h, 8h, 10h, 12h, 15h, 24h, 36h, 48h and 72h after the drug administration
Population: as for baseline characteristics
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Nintedanib: In both parts (Pilot and Main) 50 mg of nintedanib were given as a single dose on Day 1.
  In the Main part, alternatively, a single dose of 100mg could have been given. The chosen dosing scheme depended on the increase in nintedanib exposure due to ketoconazole co-administration observed in the Pilot part.
- Nintedanib + Ketoconazole: In both parts (Pilot and Main) of the study 400 mg ketoconazole were given once daily for 3 days starting on Day -2 and 50 mg nintedanib were given as a single dose 1 h after the ketoconazole administration on Day 1, with ketoconazole under steady-state conditions.
  In the Main part, alternatively, a single dose of 100mg could have been given 1 h after the ketoconazole administration or 4 h before the ketoconazole administration on Day 1. The chosen dosing scheme depended on the increase in nintedanib exposure due to ketoconazole co-administration observed in the Pilot part.
Arm/Group | Nintedanib | Nintedanib + Ketoconazole
Number analyzed (Participants) | 31 | 29
ng*h/mL | 38.6 (42.5) | 61.3 (40.4)
Statistical Analysis 1: Comparison: Nintedanib vs Nintedanib + Ketoconazole; Test type: Superiority or Other; p = 1.0000, ANOVA — p-value for ratio outside interval 0.8 - 1.25; The model includes fixed effects for sequence, period, and treatment. Subjects within sequences is included as random effect; Geometric Mean Ratio in percentage = 160.48, 90% CI 2-sided [148.245 to 173.736], Standard Deviation 17.9 — Ratio calculated as nintedanib+ketoconazole divided by nintedanib (in %). The standard deviation is actually the geometric coefficient of variation (gCV)

2. Primary Outcome: Maximum Measured Concentration (Cmax)
Description: Cmax represents the maximum concentration of nintedanib in plasma
  For this endpoint, the "measured values" show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities
Time Frame: as for outcome 1
Population: TS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Nintedanib | Nintedanib + Ketoconazole
Number analyzed (Participants) | 31 | 29
ng/mL | 4.19 (71.0) | 7.13 (44.4)
Statistical Analysis 1: Comparison: Nintedanib vs Nintedanib + Ketoconazole; Test type: Superiority or Other; p = 1.0000, ANOVA — p-value for ratio outside interval 0.8 - 1.25; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio in percentage = 179.62, 90% CI 2-sided [157.557 to 204.779], Standard Deviation 29.9 — The standard deviation is actually the gCV (in %). Ratio calculated as nintedanib+ketoconazole divided by nintedanib

3. Secondary Outcome: Area Under the Curve From 0 to the Last Quantifiable Concentration (AUC0-tz)
Description: AUC0-tz represents the area under the plasma concentration-time curve of nintedanib from time 0 to the last quantifiable nintedanib plasma concentration.
  For this endpoint, the "measured values" show inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities
Time Frame: as for outcome 1
Population: TS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Nintedanib | Nintedanib + Ketoconazole
Number analyzed (Participants) | 31 | 29
ng*h/mL | 35.7 (47.8) | 59.4 (40.8)
Statistical Analysis 1: Comparison: Nintedanib vs Nintedanib + Ketoconazole; Test type: Superiority or Other; p = 1.000, ANOVA — p-value for ratio outside interval 0.8 to 1.25; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio in percentage = 168.09, 90% CI 2-sided [155.252 to 181.981], Standard Deviation 17.9 — The standard deviation is actually the gCV. Ratio calculated as nintedanib+ketoconazole divided by nintedanib (in %)

ADVERSE EVENTS:
Time Frame: From the first trial drug administration until 18 days after the last trial drug administration, up to 32 days.
Groups:
- Ketoconazole: In both parts (Pilot and Main) of the study 400 mg ketoconazole were given once daily for 3 days starting on Day -2
Arm/Group | Ketoconazole | Nintedanib | Nintedanib + Ketoconazole
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/31 | 0/29
Other Adverse Events (participants affected / at risk) | 2/34 | 6/31 | 6/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ketoconazole (N=34) | Nintedanib (N=31) | Nintedanib + Ketoconazole (N=29)
Nasopharyngitis (Infections and infestations) | 0 | 2 | 1
Headache (Nervous system disorders) | 2 | 5 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights